CLINICAL TRIAL: NCT02176200
Title: A Randomised Open Label, Six Way, Cross-over Scintigraphic Evaluation of the Effect of Inspiratory Flow Rate on Lung and Oropharyngeal Deposition With the Respimat® Inhaler vs a Metered Dose Inhaler (HFA-MDI) Using Berodual® in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Respimat® Inhaler vs a Metered Dose Inhaler Using Berodual® in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 215.1361
Record Dates: First submitted 2014-06-24; First posted 2014-06-27 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

ARMS (2):
- Berodual® Respimat® (Experimental)
  Interventions: Drug: Berodual® Respimat®, low inspiratory flow rate; Drug: Berodual® Respimat®, medium inspiratory flow rate; Drug: Berodual® Respimat®, high inspiratory flow rate; Drug: Berodual® HFA-MDI, low inspiratory flow rate; Drug: Berodual® HFA-MDI, medium inspiratory flow rate; Drug: Berodual® HFA-MDI, high inspiratory flow rate
- Berodual® HFA-MDI (Active Comparator)
  Interventions: Drug: Berodual® Respimat®, low inspiratory flow rate; Drug: Berodual® Respimat®, medium inspiratory flow rate; Drug: Berodual® Respimat®, high inspiratory flow rate; Drug: Berodual® HFA-MDI, low inspiratory flow rate; Drug: Berodual® HFA-MDI, medium inspiratory flow rate; Drug: Berodual® HFA-MDI, high inspiratory flow rate

INTERVENTIONS:
Drug: Berodual® Respimat®, low inspiratory flow rate
Drug: Berodual® Respimat®, medium inspiratory flow rate
Drug: Berodual® Respimat®, high inspiratory flow rate
Drug: Berodual® HFA-MDI, low inspiratory flow rate
Drug: Berodual® HFA-MDI, medium inspiratory flow rate
Drug: Berodual® HFA-MDI, high inspiratory flow rate

SUMMARY:
Study to compare the lung and oropharyngeal deposition of Berodual® (fenoterol hydrobromide 50μg + ipratropium bromide 20μg /1x puff) delivered via the Respimat® inhaler and the same dose of Berodual® delivered via an hydrofluoroalkane (HFA) - metered dose inhaler (2 x puffs ) in COPD patients at different inspiratory flow rates.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have a diagnosis of COPD and must meet the following spirometric criteria:

  * Patients must have relatively stable, mild to severe airway obstruction with an forced expiratory volume in one second (FEV1) ≤70% of predicted normal and FEV1 ≤70% of forced vital capacity (FVC). Predicted normal values calculated according to evolutionary conserved chromosome segments (ECCS)
* Male or non-pregnant/non-lactating female patients aged ≥18 years
* All patients must sign an informed consent form prior to participation in the study, i.e. prior to pre-study washout of their usual pulmonary medications
* Current or ex-smokers with a smoking history of >10 pack years

Exclusion Criteria:

* Patients with significant diseases other than COPD will be excluded. A significant disease is defined as a disease which in the opinion of the investigator may either put the patient at risk because of participation in the study or a disease which may influence the results of the study or the patient's ability to participate in the study
* Patients who have frequent exacerbations which could be expected to interfere with the patient's ability to participate in the study should be excluded. The enrolment of patients who have had an exacerbation within the six weeks prior to planned study entry has to be postponed.
* Patients with clinically relevant abnormal baseline haematology, blood chemistry or urinalysis, if the abnormality defines a disease listed as an exclusion criterion will be excluded
* Patients with a recent history (i.e. six months or less) of myocardial infarction
* Patients with any unstable or life-threatening cardiac arrhythmia or who have been hospitalised for heart failure within the past year
* Patients who regularly use daytime oxygen therapy for more than 1 hour per day and in the investigator's opinion will be unable to abstain from the use of oxygen therapy
* Patients with known active tuberculosis
* Patients with a history of cancer within the last five years. Patients with treated basal cell carcinoma are allowed
* Patients with a history of life-threatening pulmonary obstruction, or a history of cystic fibrosis or bronchiectasis
* Patients who have undergone thoracotomy with pulmonary resection. Patients with a history of thoracotomy for other reasons should be evaluated as per exclusion 1
* Patients with any upper respiratory infection in the past 14 days prior to the screening visit or during the baseline period or lower respiratory tract infection within the last 3 months
* Patients who are currently in a pulmonary rehabilitation programme or who have completed a pulmonary rehabilitation programme in the six weeks prior to the screening visit
* Patients with known hypersensitivity to β2-agonists, anticholinergic drugs or any excipients of the active or placebo Berodual®
* Patients with known narrow-angle glaucoma
* Patients who are being treated with cromolyn sodium or nedocromil sodium
* Patients who are being treated with antihistamines (H1 receptor antagonists)
* Patients using oral corticosteroid medication at unstable doses (i.e. less than six weeks on a stable dose) or at doses in excess of the equivalent of 10 mg of prednisolone per day or 20 mg every other day
* Patients who are being treated with monamine oxidase inhibitors or tricyclic antidepressants
* Pregnant or nursing women or women of childbearing potential not using a medically approved means of contraception (i.e. oral or injectable eg Depo-Provera or Noristerat contraceptives, intrauterine devices, diaphragm plus spermicide or subdermal implants eg: Norplant®)
* Patients with, in the opinion of the investigator, a history of and/or active significant alcohol or drug abuse
* Patients who have taken an investigational drug within four months or six half lives (whichever is the greater) prior to screening visit and/or the administration of radiolabelled dosage forms within the three months prior to the screening visit
* Radiation exposure from clinical studies, including that from the present study and diagnostic X-rays but excluding background radiation, exceeding 5 millisievert (mSv) in the last 12 months or 10 mSv in the last five years. No patient whose occupational exposure is monitored will participate in the study

Precautions: As with other anticholinergic drugs, Berodual® should be used with caution in patients with prostatic hyperplasia or bladder neck obstruction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2003-04; Primary Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Percentage of dose in the whole lung | immediately after dosing
  disposition of aerosol via gamma scintigraphy

SECONDARY OUTCOMES:
Percentage of dose in the central lung zone | immediately after dosing
  disposition of aerosol via gamma scintigraphy
Percentage of dose in the intermediate lung zone | immediately after dosing
  disposition of aerosol via gamma scintigraphy
Percentage of dose in the peripheral lung zone | immediately after dosing
  disposition of aerosol via gamma scintigraphy
Peripheral zone/central zone deposition ratio (lung penetration index) | immediately after dosing
  disposition of aerosol via gamma scintigraphy
Percentate of dose in oropharyngeal deposition | immediately after dosing
  disposition of aerosol via gamma scintigraphy